CLINICAL TRIAL: NCT01444755
Title: Neoadjuvant Chemotherapy Versus Surgery Alone in Locally Advanced Gastric Cancer: A Randomized Controlled Study
Brief Title: The Effect of Neoadjuvant Chemotherapy on Locally Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Atilla Celik, Atilla Celik, Haydarpasa Numune Training and Research Hospital
Other Study IDs: HNEAH-01-08
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Gastric Cancer
Keywords: Locally advanced gastric cancer; neoadjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Resected stomach specimen of the patients.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1-Neoadjuvant Chemotherapy: This arm will take a neoadjuvant chemotherapy regimen previous gastrectomy operation.
- 2 Surgery: Surgery will be performed in patients of this arm.

SUMMARY:
The aim of this study is to evaluate survival benefit of a neoadjuvant chemotherapy regimen in patient with resectable locally advanced gastric cancer in comparison with surgery alone.

DETAILED DESCRIPTION:
Adenocarcinoma of the stomach ranks as the fourth most commonly diagnosed cancer and as the second leading cause of cancer-related death in the world. Radical resection with free-margin gastrectomy and extended lymphadenectomy is the preferred surgical strategy in Japan and Asian centers.

Unfortunately, only one-half of surgically treated patients with gastric cancer will achieve a complete resection without residual disease (R0) resection. Moreover, due to, the absence of routine screening programs for gastric cancer, the majority of the patients will be symptomatic at the time of diagnosis in our country.

Additionally, recent treatment strategies were focused for downsizing or decreasing to loco-regional recurrence.

In this reason, we hypothesize that preoperative chemotherapy may improve the R0 resection rate or disease free and/or overall survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of stomach
* T3 or T4
* N1 or N2
* M0
* No evidence of para-aortic or retropancreatic lymph node metastasis, peritoneal dissemination or Krukenberg tumor.
* No involvement of the esophagus with > 2cm
* An age of 18-90 years
* A Karnofsky Performance status with 60-100% or Eastern Cooperative Oncology Group (ECOG) performance status (0-2)
* No previous chemotherapy, radiotherapy for any malignancy.
* No previous surgery for gastric cancer
* No evidence obstructive or bleeding symptoms.
* Adequate renal and hepatic function
* Written informed consent

Exclusion Criteria:

* Synchronous or metachronous malignancy diagnosing within 5 year
* Pregnancy or lactation in female patients
* Any immunosuppressive condition (acquired or iatrogenic)
* Any infectious toxic or mental condition preventing neoadjuvant therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Survival | After 2 years from therapy

CONTACTS AND LOCATIONS:
Overall Officials: Atilla Celik, M.D., Principal Investigator — Haydarpasa Numune Teaching & Research Hospital, Affiliated by Ministery of Health of Turkey
Locations (1):
- Haydarpasa Numune Training and Research Hospital, Istanbul, Turkey (Türkiye)